CLINICAL TRIAL: NCT06430151
Title: Useability and Acceptability of the CUE1 Device in Older People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Alistair Mackett (Other)
Responsible Party: Sponsor-Investigator, Dr Alistair Mackett, Consultant Geriatrician, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A096551
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Useability and acceptability study of a vibrotactile stimulation device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CUE1 users (Experimental)
  Interventions: Device: CUE1

INTERVENTIONS:
Device: CUE1 — Sternal worn focused vibrotactile stimulation and cueing device

SUMMARY:
The CUE1 device is a non-invasive wearable device for people with Parkinson's Disease (PD) approved for sale in the UK. The CUE1 device utilises two established methods to improve motor symptoms in PD, namely pulsed cueing and vibrotactile stimulation. Many people with PD wish to explore non-pharmacological interventions as an adjunct to manage their motor symptom.

Study design and eligibility: This feasibility study is to establish whether the CUE1 device is a useable and acceptable device for older people with PD. 20-25 participants aged >60 years with PD will be recruited from a movement disorder service to the study.

Methodology: Participants will undertake baseline assessments of motor symptoms and quality of life with a PD nurse assessor in their own home. Following this the CUE1 device will be fitted and repeat assessments of motor symptoms will take place after 20 minutes. The participants will complete a daily diary of useability and acceptability for 4 weeks. A second visit will occur at 4 weeks with the same PD nurse assessor where the final set of motor symptom and quality of life assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals under the care of a Cambridge University Hospitals Foundation Trust movement disorder service with an established clinical diagnosis of Parkinson's disease based on the UK Brain bank criteria

Exclusion Criteria:

1. Co-existing significant neurological disorder (disabling stroke, multiple sclerosis, dementia, motor neurone disease),
2. Atypical parkinsonian disorder diagnosis (e.g. multiple systems atrophy, progressive supranuclear palsy or cortical basal degeneration syndrome)
3. co-existing physical impairment or disability causing significant mobility impairment (severe lower limb osteoarthritis)
4. trauma or pain to the sternum
5. use of other medical device e.g. pacemaker, deep brain stimulator, TENS machine etc
6. lacking capacity to consent to the study
7. Sensitivity to medical adhesives
8. Existing participant in intervention research trial

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Useability and acceptability of the CUE1 device in older people with Parkinson's disease | 4 weeks
  Participants' completion of a patient diary which will collect safety, tolerability, useability, and efficacy reports of the device over the study period. Participants will also complete a Patient Global Impression of Change (PGI-C) questionnaire at the end of the study.

SECONDARY OUTCOMES:
To undertake standardized, validated measurements of motor function with use of the CUE1 device | 4 weeks
  Completion of validated motor scores during the study period to evaluate feasibility of the data collection method for motor symptom change. Any signals of improvement in motor scores would potentially justify larger randomised controlled studies to evaluate this systematically.

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to make IPD available to other researchers